CLINICAL TRIAL: NCT06964672
Title: Advanced Imaging With Photon Counting Computed Tomography in Heart Failure Patients: a Prospective Study
Brief Title: Photon Counting Computed Tomography in Heart Failure Patients
Acronym: PCCT-HF
Status: Not yet recruiting | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: Dr Anna Mara Scandroglio (Unknown); Prof Antonio Esposito (Unknown); Prof Anna Palmisano (Unknown)
Responsible Party: Principal Investigator, Marina Pieri, MD, Università Vita-Salute San Raffaele
Other Study IDs: PCCT-HF
Record Dates: First submitted 2025-04-14; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with severe acute or chronic heart failure are increasing worldwide. Heart failure clinicians are faced daily with the need to set up short- and long- term therapeutic strategies in line with heart failure etiology and myocardial recovery chances of each patient. Current treatment strategies for severe heart failure also include mechanical circulatory support with artificial devices (such as intraaortic balloon pump, Impella, ECMO, durable left ventricular assist device), which poses specific challenges for cardiac imaging. Through its ability to directly visualize scar and evaluate its transmural extent, cardiac magnetic resonance (CMR) offers a unique advantage over other currently available imaging techniques as a central player in viability assessment in patients with coronary disease, and represents the first line technique to investigate the chances of myocardial function recovery. CMR is also an important tool to provide diagnostic data in patients with non-ischemic heart failure. Unfortunately, CMR is not feasible in many heart failure patients (for example those on MCS therapy) due to the metallic components of the mechanical devices. In these patients, the computed tomography (CT) is the alternative imaging technique to visualize cardiac structures, diagnose complications, and assess possible indications for surgical interventions. However, CT has poorer resolution and do not offer the possibility to evaluate myocardial viability in patients with contraindication to CMR. Therefore, this issue currently represents one of the major unmet needs in the clinical management of severe heart failure patients.

Recent technological advances in the field of CT imaging have nevertheless paved the way to explore new pathways of myocardial viability assessment even in patients traditionally deemed unsuitable for CMR. The introduction of photon-counting detectors, in particular, is expected to be the next major breakthrough in clinical x-ray computed tomography (CT). Photon-counting detector (PCD)-CT will overcome several shortcomings and limitations of current CT systems: it might substantially improve and expand the applicability of CT imaging by offering intrinsic spectral capabilities, increased spatial resolution, reduced electronic noise and improved image contrast. On the basis of this physical principle PCCT has the promise to improve the actual not fully satisfactory quality of scar visualization in CT images. In particular, conventional scanners are affected by a limited contrast resolution which lead to a variable and relevant rate of false negative myocardial scar-free images depending on the assessor expertise. The constant improving of CT diagnostic field have been revolutionizing the diagnostic workflow in several cardiac disease. Late contrast enhancement CT demonstrated an adequate accuracy to detect and discriminate the etiology of both ischemic and non-ischemic causes of myocardial injury compared to actual gold standard exams in patients with a troponin-positive acute chest pain syndrome. The same technique showed good sensitivity, specificity and a high negative predictive value (95%) for the identification of myocardial scars imputed to be an anatomical substrate of ventricular tachycardia with a proper concordance with electro-anatomic mapping findings (k=0.536). Finally, this enormous potential of CT implementation with the novel PCCT will provide not only the possibility to further study myocardial viability, but also is expected to be superior to standard CT exams in details definition, reduction of electronic noise and increase of spatial resolution, with consequent specific advantages in patients with heart failure, especially those with artificial devices with metallic components, in which adverse event identification and definition (such as inflow or outflow thrombosis) is complex. Thanks to these multiple diagnostic and therapeutic advantages, in combination with the availability of the PCCT device, the use of such technique is now the preferred cardiac imaging examination for the study of cardiac anatomy and function in patients with severe heart failure and a contraindication to perform the gold standard CMR. Thus, we planned a single-center observational study to asses the performance of PCCT in the identification of myocardial scars and patterns in critically ill patients with severe heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Presence of acute or chronic heart failure
* Clinical need for a CT exam with angiographic evaluation and scar imaging
* Contraindication to perform a Magnetic Resonance Imaging.
* All ages
* Signature of Informed Consent

Exclusion Criteria:

* Absence of acute or chronic heart failure
* Absence of clinical indication to a CT exam
* Contraindication to perform a CT exam.
* Pregnancy
* Refusal to provide Informed Consent to participate to the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with acute or chronic heart failure undergoing PCCT will be included in the study, upon signature of informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients with myocardial late contrast enhancement (LCE) areas | periprocedural
Identification of myocardial LCE patterns | periprocedural
  LCE patterns: endocardial, mesocardial, epicardial, transmural.
Quantification of myocardial extracellular volume (ECV) fraction. | periprocedural
  Percentage of ECV
The potential of PCCT in defining the etiology of heart failure | periprocedural
  Identification of correlation of tissue features at imaging with different diseases causing heart failure

SECONDARY OUTCOMES:
Number of patients with a PCCT detected source of infection | periprocedural
Number of patients with a PCCT detected MCS device thrombosis | periprocedural

OTHER OUTCOMES:
Residual left ventricle ejection fraction | periprocedural

REFERENCES:
- [Background] Pieri M, Ortalda A, Altizio S, Bertoglio L, Nardelli P, Fominskiy E, Lapenna E, Ajello S, Scandroglio AM. Prolonged Impella 5.0/5.5 support within different pathways of care for cardiogenic shock: the experience of a referral center. Front Cardiovasc Med. 2024 Jul 2;11:1379199. doi: 10.3389/fcvm.2024.1379199. eCollection 2024. PMID 39015682
- [Background] Barac YD, Nevo A, Schroder JN, Milano CA, Daneshmand MA. LVAD Outflow Graft Role in Pump Thrombosis. ASAIO J. 2020 Feb;66(2):128-131. doi: 10.1097/MAT.0000000000000936. PMID 30585873
- [Background] Ajello S, Pieri M, Bertoglio L, Altizio S, Nardelli P, Scandroglio AM. Extrinsic outflow graft flow obstruction in patients with HeartMate3 LVAD. Artif Organs. 2023 Apr;47(4):786-790. doi: 10.1111/aor.14450. Epub 2022 Nov 17. PMID 36385253
- [Background] Esposito A, Palmisano A, Antunes S, Maccabelli G, Colantoni C, Rancoita PMV, Baratto F, Di Serio C, Rizzo G, De Cobelli F, Della Bella P, Del Maschio A. Cardiac CT With Delayed Enhancement in the Characterization of Ventricular Tachycardia Structural Substrate: Relationship Between CT-Segmented Scar and Electro-Anatomic Mapping. JACC Cardiovasc Imaging. 2016 Jul;9(7):822-832. doi: 10.1016/j.jcmg.2015.10.024. Epub 2016 Feb 17. PMID 26897692
- [Background] Palmisano A, Vignale D, Tadic M, Moroni F, De Stefano D, Gatti M, Boccia E, Faletti R, Oppizzi M, Peretto G, Slavich M, Sala S, Montorfano M, Agricola E, Margonato A, De Cobelli F, Gentile F, Robella M, Cortese G, Esposito A. Myocardial Late Contrast Enhancement CT in Troponin-Positive Acute Chest Pain Syndrome. Radiology. 2022 Mar;302(3):545-553. doi: 10.1148/radiol.211288. Epub 2021 Dec 7. PMID 34874200
- [Background] Palmisano A, Vignale D, Benedetti G, Del Maschio A, De Cobelli F, Esposito A. Late iodine enhancement cardiac computed tomography for detection of myocardial scars: impact of experience in the clinical practice. Radiol Med. 2020 Feb;125(2):128-136. doi: 10.1007/s11547-019-01108-7. Epub 2019 Nov 29. PMID 31784926
- [Background] Sartoretti T, Wildberger JE, Flohr T, Alkadhi H. Photon-counting detector CT: early clinical experience review. Br J Radiol. 2023 Jul;96(1147):20220544. doi: 10.1259/bjr.20220544. Epub 2023 Feb 10. PMID 36744809
- [Background] Danielsson M, Persson M, Sjolin M. Photon-counting x-ray detectors for CT. Phys Med Biol. 2021 Jan 29;66(3):03TR01. doi: 10.1088/1361-6560/abc5a5. PMID 33113525
- [Background] Bock A, Estep JD. Myocardial viability: heart failure perspective. Curr Opin Cardiol. 2019 Sep;34(5):459-465. doi: 10.1097/HCO.0000000000000651. PMID 31233411
- [Background] Patel AR, Salerno M, Kwong RY, Singh A, Heydari B, Kramer CM. Stress Cardiac Magnetic Resonance Myocardial Perfusion Imaging: JACC Review Topic of the Week. J Am Coll Cardiol. 2021 Oct 19;78(16):1655-1668. doi: 10.1016/j.jacc.2021.08.022. PMID 34649703
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Al-Sabeq B, Nabi F, Shah DJ. Assessment of myocardial viability by cardiac MRI. Curr Opin Cardiol. 2019 Sep;34(5):502-509. doi: 10.1097/HCO.0000000000000656. PMID 31394561